CLINICAL TRIAL: NCT04439617
Title: Monitoring of the Mitochondrial Function of Circulating Myeloid Cells in Patients Hospitalized in the Intensive Care Unit of Dijon University Hospital
Acronym: Myelochondria
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT 2019
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Septicaemia
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis patient
  Interventions: Biological: blood examination
- Sepsis-free patient
  Interventions: Biological: blood examination

INTERVENTIONS:
Biological: blood examination — use of the remaining 1-2 ml of blood in samples taken as part of routine care to study mitochondrial function

SUMMARY:
Severe infections (sepsis) are a common cause of admission to the intensive care unit. They represent a significant health risk for patients in the short and medium term. They are particularly linked to a change in the function of immune cells. In some patients, a state of pseudo-dormancy of monocyte and macrophage-type immune cells, called immunosuppression of myeloid cells, is observed. This situation leads to a worsening of the infection, so it should be avoided because it represents a danger for the patient even when they ar receiving antibiotics. At present, these events are still very poorly understood. Research is essential to understand how this state of immunosuppression of myeloid cells is established in order to adapt existing treatments or find new ones.

Laboratory studies on animal models of septicaemia have shown that this state of immunosuppression of myeloid cells is closely linked to a change in the production of energy by myeloid cells (monocytes and macrophages). The functioning of the mitochondria ("energy factory" of the cells) in these cells is impaired. Thus, restoring mitochondrial function in myeloid cells could be a therapeutic solution against the immunosuppression of myeloid cells during severe septicaemia.

The objective of this study is to verify whether alterations in mitochondrial function in myeloid cells also occur in patients with bacterial infection compared to patients without bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult person who has given written consent (or consent obtained from a heath care proxy) hospitalized in an ICU with or without sepsis (with or without infection)

Exclusion Criteria:

* Person not affiliated or not benefiting from national health insurance
* Person under legal protection (curatorship, guardianship, safeguard of justice)
* Pregnant, parturient or breastfeeding woman
* Patient who was hospitalized within 3 months prior to inclusion for sepsis.
* Patients receiving known treatment for mitochondrial function modulation, mitochondrial biogenesis or mitophagy (chloroquine, hydroxychloroquine, rapamycin, carbamazepine, resveratrol, sildenafil).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in the ICU with or without sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Level of mitophagy in circulating monocytes | <24 hours after hospitalization in intensive care
  Measurement of mitochondrial density and PINK1 protein expression by flow cytometry in circulating monocytes (total population and subpopulation of conventional, intermediate and non-conventional monocytes (CD33, CD16 and CD14 monocyte markers)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Patoli D, Mignotte F, Deckert V, Dusuel A, Dumont A, Rieu A, Jalil A, Van Dongen K, Bourgeois T, Gautier T, Magnani C, Le Guern N, Mandard S, Bastin J, Djouadi F, Schaeffer C, Guillaumot N, Narce M, Nguyen M, Guy J, Dargent A, Quenot JP, Rialland M, Masson D, Auwerx J, Lagrost L, Thomas C. Inhibition of mitophagy drives macrophage activation and antibacterial defense during sepsis. J Clin Invest. 2020 Nov 2;130(11):5858-5874. doi: 10.1172/JCI130996. PMID 32759503